CLINICAL TRIAL: NCT05722483
Title: Intensive Virtual Treatment With Remote Abstinence Monitoring for Alcohol Use Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 055/2022
Record Dates: First submitted 2023-01-13; First posted 2023-02-10 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2023-05

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol Use Disorder; Telemedicine; Cognitive Behavioral Therapy; Dialectical Behavior Therapy
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Intensive Outpatient Program (Experimental): Participants will be treated in a 4 week program involving daily psychotherapy groups, weekly individual therapy and medication management, as well as daily breathalyzer monitoring.
  Interventions: Other: Virtual Intensive Outpatient Program

INTERVENTIONS:
Other: Virtual Intensive Outpatient Program — Components of the intervention include a cognitive behavioral therapy for alcohol use disorder group (12 sessions), a DBT skills group (12 sessions), a Health and Wellness group (8 sessions), weekly individual therapy, weekly medication management appointments, and abstinence monitoring multiple times per day using breathalyzers equipped with facial recognition and internet connectivity.

SUMMARY:
This single-arm pilot study will recruit participants with moderate to severe alcohol use disorder for a 4-week virtual intensive outpatient program (IOP). The program aims to replicate the structure and abstinence monitoring of a residential treatment program although the program is delivered entirely virtually.

DETAILED DESCRIPTION:
This pragmatic single-arm pilot study will recruit participants with moderate to severe alcohol use disorder who are seeking abstinence for a virtual intensive outpatient program (virtual IOP) The IOP will take place primarily over a 4 week period. Components of the program include a cognitive behavioral therapy for alcohol use disorder group (12 sessions), a DBT skills group (12 sessions), a Health and Wellness group (8 sessions), weekly individual therapy, weekly medication management appointments, and abstinence monitoring multiple times per day using breathalyzers equipped with facial recognition and internet connectivity. Following completion of the program, participants will complete an on-site end of treatment visit and two follow up visits at approximately day 30 and day 60 following termination of the virtual IOP. Participants will be offered the opportunity to participate in an optional weekly aftercare group for approximately 2 months after completion of the virtual IOP. Interested participants will also be able to complete optional follow-up sessions every 2 months for an additional 10 months following the end of the 60-day follow-up session.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Able to communicate and provide informed consent in English
3. Diagnosis of moderate to severe AUD, based on the Structured Clinical Interview for DSM-5, Research Version (SCID-5-RV)
4. Risky alcohol consumption, defined as > 10 drinks per week for females and > 15 drinks for males on average during the 60 days prior to the eligibility assessment.
5. Motivated to abstain from alcohol for the month-long treatment period (longer-term harm reduction goals are permitted)
6. Access to a private location from which to participate in the program for the duration of the study.
7. Able and motivated to complete all aspects of the program, including attending all virtual intensive outpatient program sessions (this includes being available for group and individual sessions throughout the day on weekdays) and completing multiple daily breathalyzer readings throughout the entire program. Individuals planning to be out of the province during the virtual intensive outpatient program will not be permitted to enroll.
8. Enrolled in the Ontario Health Insurance Plan (OHIP)

Exclusion Criteria:

1. Severe medical or psychiatric comorbidity that would prevent safe participation in the study
2. Active and severe suicidal ideation at time of eligibility assessment or suicide attempt within the past month.
3. Diagnosis of opioid use disorder or sedative use disorder within the past year based on the SCID-5 (other concurrent substance use disorders such as cannabis use disorder will not be exclusionary)
4. History of alcohol withdrawal delirium
5. Currently pregnant, breastfeeding, or intending to become pregnant or breastfeed during the study.
6. Enrollment in another study that conflicts with the procedures or scientific integrity of this study
7. Individuals planning to be out of the province during the virtual intensive outpatient program will not be permitted to enroll.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Retention in treatment | 28 Days
  Proportion of study participants that complete the entire IOP. Dropouts will include (1) individuals who miss two of the first three days of group therapy or (2) individuals who miss > 5 total days of group therapy (i.e. over 25% of the program) or (3) Participants who do not complete their breathalyzer monitoring for over 25% of the study (e.g., miss readings on > 7 days, with some exceptions). Our target retention rate to demonstrate feasibility is ≥ 50% of participants (participants who do not show up to any groups will not be included in this or other analyses).
Satisfaction with treatment as assessed by the Client Satisfaction Questionnaire-8 (CSQ-8) | 28 days
  Measures overall satisfaction with the treatment program (minimum score = 8; maximum score = 32; higher score indicates greater client satisfaction). Client satisfaction ratings in the good to excellent range (20-32) will be considered as strong evidence of acceptable levels of satisfaction with the intervention. This will be our primary measure of client satisfaction.

SECONDARY OUTCOMES:
Satisfaction with Telemedicine Delivery as Assessed by a modified version of the Telehealth Satisfaction Scale (TESS) | 28 days
  Measures satisfaction with the telehealth platform and service delivery over telehealth (minimum score = 12; maximum score = 48; higher score indicates greater satisfaction with the telemedicine platform).
Changes in Number of Abstinence Days During the IOP Assessed by the Timeline Followback Interview (TLFB) | 28 days
  Number of days in which individuals did not consume any alcohol.
Changes in Number of Binge Drinking Days During the IOP Assessed by the Timeline Followback Interview (TLFB) | 28 days
  Number of binge drinking days (4+ drinks for females, 5+ drinks for males)
Changes in Average Drinks Per Day During the IOP Assessed by the Timeline Followback Interview (TLFB) | 28 days
  Average Drinks Per Day
Change in Self-Reported Alcohol Craving During the IOP Assessed by the Penn Alcohol Craving Scale (PACS) | 28 days
  Measures craving for alcohol (minimum score = 0; maximum score = 30; higher score indicates greater levels of craving.
Change in Quality of Life during the IOP Assessed Using the Abbreviated World Health Organization Quality of Life Scale (WHOQOL-BREF) | 28 days
  Measures quality of life (scores are transformed to 0-100; higher scores indicate higher quality of life).
Change in Depressive Symptoms during the IOP Assessed Using the Patient Health Questionnaire-9 (PHQ-9) | 28 days
  Measures depressive symptoms (minimum score = 0; maximum score = 27; higher scores indicate higher levels of depressive symptoms).
Change in Anxiety Symptoms during the IOP Assessed Using the Generalized Anxiety Disorder-7 (GAD-7) | 28 days
  Measures generalized anxiety (Minimum score = 0; maximum score = 21; higher scores indicate higher levels of anxiety)
Change in Sleep during the IOP Assessed Using the Pittsburgh Sleep Quality Index (PSQI) | 28 days
  Measures quality of sleep (minimum score = 0; maximum score = 21; higher scores indicate lower quality of sleep).
Change in Emotion Regulation During the IOP Assessed Using the Difficulties in Emotion Regulation Scale (DERS) | 28 days
  Measures difficulties in emotion regulation (minimum score = 36; maximum score = 180; higher scores indicate more difficulties in emotion regulation)
Change in Emotion Regulation During the IOP Assessed Using the Emotion Regulation Questionnaire (ERQ) | 28 days
  Measures cognitive reappraisal (minimum score = 6; maximum score = 42; higher score indicates more frequent use of reappraisal) and expressive suppression (minimum score = 4; maximum score = 28; higher scores indicate more frequent use of suppression).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Sloan, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No